CLINICAL TRIAL: NCT02358785
Title: Evaluation of a Powered Stapler System on Surgical Interventions Required During Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC-14-005
Record Dates: First submitted 2015-01-30; First posted 2015-02-09 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: ECHELON FLEX™ Powered Plus Stapler — ECHELON FLEX™ Powered Plus Stapler using ENDOPATH ECHELON™ Reloads with Gripping Surface Technology (GST). The combination of stapler plus reload is referred to as the ECHELON FLEX™ GST System.

SUMMARY:
This study will provide clinical data in an observational setting. Individuals undergoing LSG, and who meet study entry criteria, may be enrolled. LSG procedures will be performed according to institutional standard-of-care (SOC) using the study stapler. All study subjects will be followed for approximately 4 weeks for safety and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for laparoscopic sleeve gastrectomy;
* Subject meets NIH weight loss surgical criteria;
* BMI ≤ 60 kg/m2;
* Willing to give consent and comply with study-related evaluations; and
* At least 18 years of age

Exclusion Criteria:

* Previous bariatric procedures, including gastric banding;
* Prior gastric surgery;
* Scheduled concurrent surgical procedure (hiatal hernia repair, cholecystectomy allowed);
* Pregnancy;
* Known or suspected uncontrolled bleeding disorders;
* History of chronic steroid use;
* Patients who have undergone significant upper GI surgery leading to adhesion; formation, as determined by the Principal Investigator;
* Physical or psychological condition which would impair study participation;
* The patient is judged unsuitable for study participation by the Investigator for any other reason; or
* Unable or unwilling to attend follow-up visits and examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals scheduled for laparoscopic sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Surgical interventions (type, quantity, frequency, rationale) required during LSG | Intraoperative

SECONDARY OUTCOMES:
Procedure duration | Up to one day
Length of stay | Up to 4 weeks
Estimated blood loss | up to one day

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Fernandez, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Surgical Specialists of Louisiana, Metairie, Louisiana
  - Carolinas Weight Management, Charlotte, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Greenville Health System, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
via publication